CLINICAL TRIAL: NCT03214289
Title: Fecal Microbiota Transplantation for Treatment of Steroid Resistant and Steroid Dependent Gut Acute Graft Versus Host Disease- a Pilot Study
Brief Title: Fecal Microbiota Transplantation for Steroid Resistant and Steroid Dependent Gut Acute Graft Versus Host Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Shouval Roni, Principal Investigator, Hematology and BMT Division, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3822-16-SMC; 3822-16-SMC (Other: Sheba Medical Center, Tel-HaShomer, Israel)
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Stem Cell Transplant Complications; Graft Versus Host Disease, Acute; Fecal Microbiota Transplantation
Keywords: Fecal Microbiota Transplantation; Intestinal Acute Graft Versus Host Disease; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (FMT) (Experimental): Participants will receive a single dose of oral FMT, which is 15 capsules per day for 2 consecutive days (total of 30 capsules). All capsules administered to a participant are from the same unrelated donor. Participants will be asked to fast for 4 hours prior to and 1 hour following capsule intake. Participants will be asked to drink at least 360cc of water during administration.
  Treatment will be administered on an inpatient basis. In patients with no/partial response, the FMT may be repeated from the same or a different donor.
  Subjects receiving any amount of the FMT capsules will be followed for at least 6 months.Stool and blood samples will be serially collected.
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Thirty fecal microbiota capsules produced from a single healthy donor, unrelated to the participant.

SUMMARY:
The investigators hypothesize that perturbations in the intestinal microbiota following allogeneic hematopoietic stem cell transplantation (HSCT) are essential for the development and propagation of acute graft-versus-host disease. Therefore, modification of HSCT recipients' gut microbiota using fecal transplantation from a healthy donor could be used to treat gut acute GVHD.

The study evaluates safety and feasibility of fecal microbiota transplantation with frozen capsules from healthy donors for the treatment of steroid resistant or steroid dependent acute graft-versus-host disease of the gut.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18 to 75 years) who underwent allogeneic hematopoietic stem cell transplantation (HSCT) and developed gut acute Graft-versus-Host Disease (aGvHD).
* Participants have steroid-resistant or steroid-dependent gut aGvHD.
* Steroid resistant gut aGvHD is defined as cases in which gastrointestinal symptoms do not improve within 7 days after initial steroid therapy (≥1 mg/kg of methylprednisolone) or clear progression after 5 days.)
* Steroid-dependent gut aGVHD is defined as cases in which reduction of steroid dose was not possible due to exacerbation of gastrointestinal symptoms.
* Participants may have undergone allogeneic HSCT for any diagnosis at any time prior to developing aGvHD, and are not restricted to any specific conditioning regimen or by the subsequent administration of donor lymphocyte infusion.
* Participants should be able to give informed consent.

Exclusion Criteria:

* Participants may not have gut aGvHD which permits the tapering of steroid dose.
* Participants may not have ongoing, uncontrolled infection (i.e. unresolved bacteremia, uncontrolled CMV infection).
* Participants may not have ongoing enteritis primarily caused by enteropathy other than gut GvHD, excluding resistant clostridium difficile infection.
* Participants may not have acute neutrophil count < 500 cells/µL.
* Participants may not have toxic megacolon
* Participants may not have active gastrointestinal bleeding.
* Participants may not be pregnant or lactating.
* Participants may not be unable to swallow pills.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-07-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | 28 days following FMT.
  Participants will be evaluated for serious adverse events (SAEs) relating to FMT occurring within 28 days following transplantation. SAEs are defined as any adverse experience occurring during or after FMT that results in any of the following outcomes: death, life-threatening experience, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity or an important medical event events

SECONDARY OUTCOMES:
Non-serious adverse events | 28 days following FMT.
  Participants will be evaluated for non-serious adverse events relating to FMT within 28 days following transplantation. Non-serious adverse events are defined as diarrhea, nausea and vomiting, fatigue and malaise, headache, and distension/bloating/abdominal discomfort/pain
Gut acute Graft-versus-Host Disease (aGvHD) response. | up to 28 days following FMT.
  Participants will be evaluated on days 7 and 28 following transplantation for response to therapy.
  Response criteria for steroid-resistant patients is as follows:
  * Complete response: resolution of all gastrointestinal signs and symptoms
  * Partial response: decrease in severity of gut GVHD by at least one stage
  * Progression: Progressive worsening of gut GVHD
  * No change: No significant change in gut GVHD
  Response criteria for steroid-dependent patients is as follows:
  * Complete response: reduction of the steroid dose to 5 mg or less of prednisone (or a steroid equivalent) per day.
  * Partial response: a reduction of ≥40% in the dose of steroid
  * Progression: an increase of >=10% in the steroid dose
  * No change: any other option
aGvHD severity | up to 28 days following FMT.
  Participants will be evaluated on days 7 and 28 following transplantation for severity of aGvHD.
  aGVHD severity is graded by the International Bone Marrow Transplant Registry Severity Index grading system
Reduction in the dose of steroids. | up to 28 days following FMT.
  The dose of methylprednisolone, or an equivalent GCS, will be evaluated on day 7, and 28. The change in the dose at day 28, adjusted to the type of GCS used.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Shouval, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No